CLINICAL TRIAL: NCT06221423
Title: A Single-center, Prospective Cohort Study of Fruquintinib Combined With TAS-102 in Refractory Metastatic Colorectal Cancer
Brief Title: Fruquintinib Combined With TAS-102 in Refractory Metastatic Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Director of Colorectal Surgery, Fudan University
Other Study IDs: Fru plus TAS-102 in mCRC
Record Dates: First submitted 2023-12-27; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer; Metastatic Colorectal Cancer; Refractory Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fru plus TAS-102: mCRC patients receiveing Fruquintinib combined with TAS-102 in third- or late- line
  Interventions: Drug: Fruquintinib Combined With TAS-102

INTERVENTIONS:
Drug: Fruquintinib Combined With TAS-102 — Fruquintinib Combined With TAS-102

SUMMARY:
Fruquintinib, as a standard treatment for refractory metastatic colorectal cancer (mCRC), has attracted increasing research efforts to explore its innovative strategies in combination with immunotherapy and chemotherapy because of its multi-target mechanism which enhances the sensitivity of the immune system and chemotherapy, aiming to further improve the survival benefits for mCRC patients. Trifluridine/tipiracil (TAS-102) is also a standard treatment for mCRC. This study aims to investigate the safety and effectiveness of the combined use of these two drugs in mCRC.

ELIGIBILITY:
Inclusion Criteria:

* Histology-confirmed metastatic CRC (mCRC)
* Disease progression on standard therapy with at least two lines of chemotherapy, including fluorouracil, oxaliplatin, and irinotecan with or without biologics such as bevacizumab and cetuximab
* Fruquintinib administered as salvage treatment
* Age: 18-75 years old
* Informed consent

Exclusion Criteria:

* Liver or kidney dysfunction, or other conditions unsuitable for chemotherapy
* Fruquintinib and/or TAS-102 administration as second-line treatment
* Drug administration stopped after less than two cycles

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with refractory metastatic colorectal cancer who have undergone third-line or later treatment with a combination of fruquintinib and TAS-102.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | 3 years
  PFS was calculated from the date of fruquintinib administration to the first observation of disease progression or death.
Overall Survival (OS) | 3 years
  OS was defined as the time from fruquintinib administration to death.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, Principal Investigator — Department of Colorectal Surgery, Zhongshan Hospital, Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided